CLINICAL TRIAL: NCT04296149
Title: Studio Esplorativo Monocentrico Non Controllato, in Aperto, Volto a Sviluppare e Valutare l'Applicazione di Una Tecnica Innovativa di Rimozione Radioguidata Dei Tumori Neuroendocrini Gastro-entero-pancreatici
Brief Title: Beta- Probe and Surgery in GEP NET: Evaluation of a New Probe
Acronym: RADIONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 0388
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Tumors
Keywords: beta- probe; radioguided surgery
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 90Y-octreotide, DOTA-Tyr(3)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Y-90-DOTATOC (Experimental): Patients affected by Small Intestine neuroendocrine tumors
  Interventions: Drug: Y90-DOTA-Tyr3-Octreotide

INTERVENTIONS:
Drug: Y90-DOTA-Tyr3-Octreotide — Patients enrolled for surgery will receive a small amount of Y-90-DOTATOC, in order to check beta- radioactivity by the probe
  Other Names: Beta- emetting radioisotope

SUMMARY:
Radioguided surgery (RGS) with beta- radioisotopes is a novel approach focused on developing a new probe which, detecting electrons and operating with low background, provides a clearer delineation of the margins of lesions with low radiation exposition for surgeons.

To validate this procedure, ex vivo specimens of tumours expressing somatostatin receptors, as small-intestine neuroendocrine (SI-NET), will be tested

DETAILED DESCRIPTION:
Small Intestinal neuroendocrine patients, with a positive Ga-68-DOTATOC PET/CT, will receive a small amount of beta- radiopharmaceutical (Y-90-DOTATOC), and then operated, as clinical indicated.

Tissue samples will be tested ex-vivo with a beta-probe prototype

ELIGIBILITY:
Inclusion Criteria:

* SI NET patients, Ga-68-DOTATOC PET/CT positive, proposed for surgery

Exclusion Criteria:

* negative PET/CT; pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensitivity of a beta- probe | 2 years
  after receiving a small amount of radioactivity, patients will be operated and an evaluation of radioactivity on surgical specimens will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Chiara Maria Grana, Milan, Italy